CLINICAL TRIAL: NCT03425123
Title: Endodontic Regenerative Procedure for Immature Non-vital Teeth
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not started due to the lack of funding.
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-37079
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Tooth, Nonvital
Keywords: Regenerative endodontic procedure (REP); Mineral Trioxide Aggregate (MTA) apexification; Calcium Hydroxide -Ca(OH)2; Permanent non-vital tooth; Children 7-18 years of age
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REP Group (Experimental): All participants in this single arm study will receive Regenerative Endodontic Procedure (REP). It regenerates the root tip on recently erupted permanent teeth that did not complete root development due to pulp infection and necrosis by allowing cells to migrate from the surrounding periapical tissue and enter the pulp space. Cells contained within the intentional bleeding create at the root tip help in root completion as well as increasing the thickness of the canal walls over up to two years following the procedure.
  Interventions: Other: Regenerative Endodontic Procedure (REP)

INTERVENTIONS:
Other: Regenerative Endodontic Procedure (REP) — Regenerative Endodontic Procedure (REP) involves disinfection of the root canal with the use of acombination of three antibiotics including ciprofloxacin, metronidazole, minocycline. At the second visit, the patient is evaluated for resolution of signs or symptoms of an acute infection and if none then bleeding is induced, the site covered with a plug and the patient is evaluated at follow up.

SUMMARY:
In this clinical trial the investigators will evaluate an alternate treatment option, which was developed for teeth with incomplete roots, called Regenerative Endodontic Procedure (REP). This treatment works by harnessing the blood clot formed within the root canal from tissues surrounding the root as a scaffold for stem cells. These cells could help to increase the thickness and length of the root canal walls resulting in root end maturation.

Results from the 50 participants who will receive the REP treatment will be compared with findings with historical data.

DETAILED DESCRIPTION:
All participants will be prospectively assigned to the REP treatment group. Results from the treatment group will be compared to historical controls of all subjects treated by Ca(OH)2 or MTA apexification in the last 10 years (2007-2017) at the Boston University Henry M Goldman School of Dental Medicine.

All materials used in this protocol are FDA approved and commercially available for similar applications. This study does not seek a new use or application of any materials, instead recommendations of the American Association of Endodontists (AAE) will be followed to evaluate outcomes associated with the REP compare to the standard of care Ca(OH)2 or MTA apexification.

The overall objective for this research is the elimination of any clinical symptoms and the evidence of bony healing as examined by radiographs.

Other objectives include increased root wall thickness and/or increased root length and positive response to vitality testing, which if achieved, could indicate a more organized vital pulp tissue.

ELIGIBILITY:
Inclusion Criteria:

Subjects followed prospectively

* 7-18 years old
* salvageable permanent non-vital tooth with immature apex whether anterior or posterior
* receiving dental care at the Henry M. Goldman School of Dentistry Historical controls
* 7-18 year old
* salvageable permanent non-vital tooth with immature apex whether anterior or posterior
* received care and has accessible records at the Henry M. Goldman School of Dentistry
* had either the Calcium hydroxide apexification or MTA apexification between 2007 and 2017

Exclusion Criteria:

* allergic to medications necessary to complete procedure
* health status not in: a) ASA-1 no organic pathology or patients in whom the pathological process is localized and does not cause any systemic disturbance or abnormality; nor b) ASA 2 A moderate but definite systemic disturbance, caused either by the condition that is to be treated or surgical intervention or which is caused by other existing pathological processes
* history of dental trauma within 6 months due to possibility of internal and external root resorption.
* if tooth pulp space is needed for post/core final restoration
* pregnancy in female subjects

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
periradicular bone healing | 24 months
  Bone healing will be determined by calculating the difference in the bone thickness in millimeters comparing baseline to 24 months on radiographs
periradicular bone infection | 1-4 weeks after first visit
  Assess and document any signs/symptoms of infection at the second visit

SECONDARY OUTCOMES:
tooth root thickness at 12 months | 12 months
  The tooth root thickness will be measured in millimeters, comparing the pre-procedure radiographs and Cone-Beam-Computed Tomography scans (CBCT) to radiographs and CBCT at 12 months
tooth root thickness at 24 months | 24 months
  The tooth root thickness will be measured in millimeters, comparing the pre-procedure radiographs and Cone-Beam-Computed Tomography scans (CBCT) to radiographs and CBCT at 24 months
tooth root length at 12 months | 12 months
  The tooth root length will be measured in millimeters, comparing the pre-procedure radiographs and Cone-Beam-Computed Tomography scans (CBCT) to radiographs and CBCT at 12 months
tooth root length at 24 months | 24 months
  The tooth root length will be measured in millimeters, comparing the pre-procedure radiographs and Cone-Beam-Computed Tomography scans (CBCT) to radiographs and CBCT at 24 months
tooth vitality at 12 months | 12 months
  A pain response to hot/cold and electrical pulp tester will be done to test the vitality of the tooth pulp at 12 months
tooth vitality at 24 months | 24 months
  A pain response to hot/cold and electrical pulp tester will be done to test the vitality of the tooth pulp at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sami Chogle, BDS DMD MSD, Study Director — Henry M Goldman School of Dental Medicine
Locations (1):
- Henry M Goldman School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No